CLINICAL TRIAL: NCT06207448
Title: Deep Infiltrating Endometriosis : Laparoscopic Nerve-sparing Surgery and Use of Neutral Argon Plasma
Acronym: DIE
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8501
Record Dates: First submitted 2023-12-11; First posted 2024-01-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis Ovary
Keywords: Endometriosis Ovary; Laparoscopic Surgery; Laparoscopic Surgical Procedure; Schwanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medical treatment of endometriosis has a suspensive and sometimes incomplete effect on the symptoms, making surgical treatment necessary. The aim of surgical treatment of deep endometriosis is to restore normal anatomy and functional integrity. Resection of deep endometriosis lesions is recommended to relieve pain, gynecological and digestive symptoms, but rarely urinary disorders. Nerve-sparing surgery, when feasible, reduces post-operative dysuria by sparing the lower hypogastric plexus.

The major limitations of these surgical procedures are the experience of the surgeon and the extent of the disease. Acquiring the surgical techniques and skills necessary to carry out these types of procedures is essential to providing optimal patient care.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (≥18 years old)
* Patient who benefited from treatment by nerve-sparing surgery and the use of neutral argon plasma in the context of symptomatic deep pelvic endometriosis at the Strasbourg University Hospital during 2021
* Patient who did not express, after information, the reuse of her data for the purposes of this research.

Exclusion Criteria:

* Patient who expressed her opposition to participating in the study
* Patient under legal protection, under guardianship or under curatorship

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult woman (≥18 years old) who benefited from treatment by nerve-sparing surgery and the use of neutral argon plasma in the context of symptomatic deep pelvic endometriosis at the Strasbourg University Hospital during 2021
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
To retrospectively describe the minimally invasive management of deep pelvic endometriosis using nerve-sparing surgery and the use of neutral argon plasma for extensive endometriotic lesions by laparoscopy | up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie Obstétrique - CHU de Strasbourg - France, Strasbourg, France